CLINICAL TRIAL: NCT03197623
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Single and Multiple Ascending Dose Study of the Safety and Tolerability of Intravenous LLP2A-Alendronate in Adult Men and Women With Osteopenia Secondary to Glucocorticoids
Brief Title: Safety and Tolerability of Intravenous LLP2A-Alendronate for Osteopenia Secondary to Glucocorticoids
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nancy E. Lane, MD (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor-Investigator, Nancy E. Lane, MD, Professor, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 20161825; LLP2A-001 (Other: UC Davis)
Record Dates: First submitted 2017-04-19; First posted 2017-06-23 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Osteopenia; Osteoporosis; Osteonecrosis
Keywords: Glucocorticoids
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis; Osteonecrosis

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled Single and Multiple Ascending Dose Study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LLP2A-ALENDRONATE (Experimental): 50, 150, 400, 750 or 1200 μg/kg or placebo given as a one time intravenous administration over 120 minutes.
  Interventions: Drug: LLP2A-ALENDRONATE
- Placebo (Placebo Comparator): Placebo given as a one time intravenous administration over 120 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LLP2A-ALENDRONATE — A small molecule, LLP2A-Ale that directs endogenous mesenchymal stem cells (MSCs), the cells that have the potential to grow bone tissue, to the bone surface to form new bone. Single administration of LLP2A-Ale given intravenously over 120 minutes.
  Other Names: LLP2A-Ale
  Arms: LLP2A-ALENDRONATE
Drug: Placebo — Placebo, one time single administration given intravenously over 120 minutes.
  Arms: Placebo

SUMMARY:
A Phase 1 Randomized, Double-Blind, Placebo-Controlled Single and Multiple Ascending Dose Study of the Safety and Tolerability of Intravenous LLP2A-Alendronate in Adult Men and Women with Osteopenia Secondary to Corticosteroids

DETAILED DESCRIPTION:
The study is designed to evaluate safety and tolerability of LLP2A-Ale beginning with a single ascending dose (SAD) cohort followed by multiple ascending dose (MAD) cohorts with matching placebo in each cohort. The population in this study includes patients with low bone density (osteopenia with a T score ≤ -1.0) in the femoral neck, total hip or lumbosacral spine who are taking Corticosteroids. Up to 59 patients will be enrolled, 32 in the SAD and 27 in the MAD.

LLP2A-Ale is a novel anabolic agent. It appears that LLP2A-Ale may have utility in a variety of conditions where new bone formation is required. Non-traumatic osteonecrosis (ON) has been selected as the first indication for LLP2A-Ale because of the high unmet need, absence of treatments besides surgical joint replacement, and the clear need to attract and stimulate differentiation of stem cells into the region of necrotic bone. However, osteonecrosis is a rare, sporadic disease. Therefore, the Phase 1 study is being performed in people at risk for osteonecrosis, as a population representative of people with osteonecrosis, who will be the participants in any subsequent Phase 2 and 3 studies.

Non-traumatic ON may also be caused by a variety of underlying medical conditions. Glucocorticoid use, alcohol, and smoking contribute to up to 80% of cases of nontraumatic ON. The relationship to GC is the strongest in people receiving relatively long term therapy, with risk increasing with cumulative exposure over three or more months. Vasculitis from autoimmune diseases predisposes to ON and ON is particularly associated with Systemic Lupus Erythematous (SLE), possibly due to coexistence of vasculitis and chronic GC treatment. In different series, symptomatic ON is reported in about 5-30% of SLE patients. Because many foci of ON are asymptomatic, rates based on MRI surveillance are higher, in the range of 30 - 50%, and often are multifocal. Because of the particularly high incidence of ON in SLE we anticipate that SLE patients will be a significant component of the population in later trials. Therefore investigators in this Phase 1 trial include rheumatologists in order to increase the likelihood of inclusion of lupus patients in this first study.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be included in the study.

1. 20 - 85 years old
2. Receiving 5 - 40 mg/day prednisone, or equivalent of another GC (methylprednisolone 4 mg/day, or prednisone 10 mg every other day) for a minimum of 4 consecutive weeks prior to enrollment
3. Anticipated to continue to receive at least 5 mg/day prednisone or equivalent throughout study participation
4. T score ≤ -1.0 in the femoral neck or total hip or lumbosacral spine. Only one result from one of these locations that is ≤ -1.0 is required. For screening DXA, a DXA completed within 6 months of screening may be used; otherwise DXA must be completed within 4 weeks of screening visit.
5. Must be ambulatory and able to attend all appointments
6. Women must agree to use one of the following methods of birth control for the duration of the clinical trial: systemic hormonal contraceptive (oral, injected, transdermal), intrauterine device, double barrier (e.g., cervical cap or diaphragm with condom or spermicide). Men with female partners must agree to use double barrier contraception, unless their partner is using systemic hormonal contraceptives or has an intrauterine device.
7. In the opinion of the investigator, the concurrent medical conditions of the study subject are stable
8. Subject undergoing PET/CT scans must have the ability to lay motionless for up to 30-45 minutes
9. Anticipated to continue to receive all chronic medications without dose changes throughout study participation
10. Subjects undergoing PET/CT scans must have the ability to lay motionless for up to 30-45 minutes

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. Weight greater than the limit of the DXA table at the clinical site
2. History or concurrent conditions that might place the subject at increased risk, such as renal insufficiency (CKD 4 or 5), glomerulonephritis, atypical infections due to impaired immunity, hypersensitivity to multiple IV medications
3. History of or concurrent presence of medical conditions which might interfere with ability to participate for the duration of the study, such as clinically significant cardiovascular disease, uncontrollable hypertension, uncontrolled asthma, symptomatic pulmonary fibrosis, recent GI bleeding requiring transfusion, psychosis, substance abuse or hospital admission within 6 months of enrollment (except for elective procedures)
4. Prior use or current need for prohibited concomitant medications
5. Rheumatic disease with clinically significant renal or central nervous system involvement
6. History of deep vein thrombosis (DVT) along with taking any prophylaxis/treatment that occurred within the last 5 years
7. History of clinically significant atrial fibrillation and/or taking medications for its treatment and prevention
8. Unable or unwilling to comply with restrictions on alcohol 9. Previous hypersensitivity to alendronate

10. Any of the following on Screening laboratory tests:

1. Total calcium values outside the normal range (corrected if albumin < lower limit of normal (LLN))
2. Phosphate level < LLN
3. 25-hydroxyvitamin D (25-OH Vitamin D) below 10ng/mL
4. TSH > upper limit of normal (ULN)
5. Hepatic enzymes (ALT, AST, GGT) > 1.5 X ULN
6. Creatinine clearance (eGRF) <35 mL/min/1.73 m2 using the Modification of Diet in Renal Disease (MDRD) formula
7. Hemoglobin <10 g/dL
8. Positive serology for HIV, Hepatitis B or C
9. Positive pregnancy test
10. Prolonged QTc interval (QTcF (Fredericia) of > 450 msec for men, > 470 msec for women)
11. Any other clinically significant laboratory value as judged by the investigator 11. Subject cannot enroll in MAD part of study until after 60 days of completing SAD part of study 12. Subjects undergoing PET/CT scans must not be breast-feeding 13. History of hypersensitivity to fluoride

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Dose limiting Adverse events | Duration of the Study, average of 4 years
  Incidence of dose limiting or intolerable treatment related adverse events (AEs) including A serious drug-related adverse event in ≥ 1 subject receiving LLP2A-Ale and/or Severe drug related adverse events in ≥ 2 subjects receiving LLP2A-Ale

SECONDARY OUTCOMES:
Severe infusion reactions | Duration of the study, average of 4 years
  Fever, myalgia, nausea/vomit, headache, flu like symptoms in ≥ 2 subjects receiving LLP2A-Ale
Grade 2 elevated creatinine | Duration of the study, average of 4 years
  serum creatinine greater than 1.5 - 3.0 x baseline; greater than 1.5 - 3.0 x upper limit of normal (CTCAE v4.0) in ≥ 1 patient.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Lane, MD, Principal Investigator — UC Davis Health; Nancy E Lane, MD, Study Director — UC Davis Health
Locations (4):
- United States (4):
  - West Coast Clinical Trials (WCCT), Cypress, California
  - Diablo Clinical Research, Walnut Creek, California
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided